CLINICAL TRIAL: NCT05262296
Title: A Single Blinded Randomised Controlled Trial Comparing the Ergonomics of Laparoscopic and Versius Robotic Assisted Colorectal Surgery
Brief Title: Versius or Laparoscopic Colorectal Cancer and Non-cancer Operation Outcomes
Acronym: VOLCANO
Status: Completed | Type: Observational
Sponsor: Joanne Turner (Other Government)
Responsible Party: Sponsor-Investigator, Joanne Turner, Academic Research Coordinator, Milton Keynes University Hospital NHS Foundation Trust
Organization: Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Other Study IDs: MKUH-RD-020
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Disorders
Keywords: robotic surgery; laparoscopic surgery; ergonomics; Versius

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic Surgeon: This cohort of participants will have their procedure completed by a human surgeon.
  Interventions: Procedure: Laparoscopic Surgeon
- Robotic Arm: This cohort of participants will have their procedure completed by the Versius Surgical Robotic System
  Interventions: Procedure: Robotic Arm

INTERVENTIONS:
Procedure: Laparoscopic Surgeon — Laparoscopic Arm This cohort of participants will have their procedure completed by a human surgeon.
  Groups: Laparoscopic Surgeon
Procedure: Robotic Arm — This cohort of participants will have their procedure completed by the Versius Surgical Robotic System.
  Groups: Robotic Arm

SUMMARY:
This is a study comparing major bowel surgery done via conventional keyhole (laparoscopic) surgery with robotic assisted keyhole surgery, using the Versius robotic system. Our main objective is to assess the physical strain of both types of surgery on the operating surgeon, but we will also collect data on the patient outcomes and teamwork. This results from this study will be used to guide the design of a larger scale trial in future.

DETAILED DESCRIPTION:
This study has been designed to assess the ergonomics of Versius® assisted surgery in comparison with laparoscopic surgery in the management of major colorectal resection. The study will randomise 60 patients who require removal of either part or all of the colon or rectum and have been deemed suitable for a minimally invasive approach, as management of either benign or malignant colorectal pathology.

Patients will be randomised to receive either laparoscopic or Versius® robotic assisted surgery but will be informed that it will be attempted via a minimally invasive approach that could include either of these two subtypes of minimally invasive surgery. The randomisation will occur on a 2:1 basis, with 2 patients allocated to the robotic arm for every 1 patient allocated to the laparoscopic arm. Laparoscopic surgery is already a well-established technique, and therefore the study team believe more valuable data about the outcomes of robotic surgery will be obtained with this randomisation ratio given that no prior studies have been undertaken using this robotic platform.

All surgeons in the study will be required to have been involved in at least 20 cases performed using the relevant modality, whether for the robotic or laparoscopic cohorts.

Data will be collected at four key timepoints; recruitment, intraoperatively, at discharge and again at 28 days following intervention. Feasibility outcomes will include willingness to be recruited to study (acceptability), willingness for patient to undergo desired randomised operative approach (acceptability/concordance), withdrawal of patients (non-concordance), study retention (retention rates), and the usefulness and limitations of outcome measures.

The study outcomes examined will relate to the patient, the surgeon performing the procedure, and also cost of the procedure. Surgeon specific outcomes will include measurement of physical and mental strain encountered during the procedures as assessed by the REBA and NASA-TLX scales. Patient specific outcomes will include quality of life analysis (EQ-5D-5L and MFSI-SF scores), hospital length of stay duration, post-operative complications, conversion to open surgery and pain scores. Assessment of intraoperative theatre team communication will be measured using the Oxford NOTECHS II scale which is a modification of a scale originally used in aviation, but adapted and widely validated for use in surgical contexts. The cost of equipment used during the procedure, the cost of theatre utilisation, and the total cost of the inpatient admission will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Need for colonic or rectal resectional surgery
* Deemed suitable for minimally invasive surgery

Exclusion Criteria:

* Patients who are unable to consent
* Prisoners
* Patients in need of emergency surgery
* High likelihood of treatment delays caused by randomisation process (e.g. due to lack of operative capacity for one approach)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who require surgery to remove part or all of the colon or rectum will be approached to participate in the trial.
  In this trial, all patients will be only be considered if deemed suitable for surgery via a minimally invasive approach
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
To compare the operating surgeon ergonomics (physical strain) of laparoscopic and Versius® robotic assisted surgery | Length of the procedure expected to be between 1-4 hours
  body position (physical strain) and cognitive workload (mental strain) assessed using the REBA score

SECONDARY OUTCOMES:
Measurement of the rate of participant recruitment | Through study completion, an average of 1 year.
  Measure the number of participants recruited over the length of time. The units of measurement will be presented on a scale of number of participants over a predetermined length of time
Measurement of drop-out (withdrawal) rate of participants | Assessed from Day 1 (Randomisation) to date of withdrawal
  Measure the number of participants who withdrawal (drop out) from the trial. The units of measurement will be presented on a scale of numbers of withdrawals versus time.
Measurement of the unblinding rate of participants | Through study completion, an average of 1 year.
  Measure the number of participants where the treatment is unblinded during the trial. This is measured by the number of participants over the length of time who's treatment is unblinded.
Mental strain of surgeon | 30 minutes maximum completion time per surgeon
  To compare the operating surgeon mental strain of each approach using the NASA-Task Load Index score
Health Economics | Procedure and recovery inpatient stay per participant expected to be between 1-3 days
  Explore health economic aspects of each approach via calculation of the entire hospital episode and individual operation (including fixed costs and instrument costs) comparing the cost for cohort using the Versus Surgical Robot versus the human surgeon.
Satisfaction with life scale | Assessed on Day 28
  Quality of life units completion of EQ-5D-5L questionnaire post operatively on day 28. Total scores used not sub scales to be reported.
Quality of life scale | Assessed on Day 28
  Quality of life units completion of MFSI-SF questionnaire post operatively on day 28. Total scores used not sub scales to be reported.
.Pain Scores | Days 1, 2, 3 and 28
  Using a uni-dimensional pain score measurement examining the change from baseline.
Communication | 1-4 hours expected for the duration of the procedure
  To compare differences in in-theatre communication assessed from audiovisual footage, using the Oxford NOTECHS II score.

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Keeler, Principal Investigator — Consultant Colorectal Surgeon
Locations (1):
- Milton Keynes University Hospital, Milton Keynes, Bucks, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dixon F, Vitish-Sharma P, Khanna A, Keeler BD; VOLCANO Trial Group. Robotic assisted surgery reduces ergonomic risk during minimally invasive colorectal resection: the VOLCANO randomised controlled trial. Langenbecks Arch Surg. 2024 Apr 27;409(1):142. doi: 10.1007/s00423-024-03322-y. PMID 38676748